CLINICAL TRIAL: NCT03219983
Title: Pain Management After Total Shoulder Arthroplasty: Continuous Interscalene Block Versus Local Tissue Infiltration With Liposomal Bupivacaine
Brief Title: Pain Management After Total Shoulder Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: The Christ Hospital (Other)
Responsible Party: Principal Investigator, Dr. Paul Favorito, Principal Investigator, The Christ Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Total Shoulder
Record Dates: First submitted 2017-02-28; First posted 2017-07-18 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-07

CONDITIONS: Glenohumeral Arthritis; Total Shoulder Arthroplasty
Keywords: interscalene block; liposomal bupivacaine
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Interscalene Block (Active Comparator): Ultrasound guided interscalene catheter will be placed and a 30 ml .5% ropivacaine will be given pre-operatively. Upon arrival to the Post-Operative Care Unit a continuous infusion of .5% ropivacaine will be started at 8ml/hr and increased by 2ml/hr every 15 minutes for pain score > 4 with a maximum rate of 14ml/hr. Infusion will be delivered by ON-Q Select-a-Flow pump (volume 750ml)
  Interventions: Drug: Ropivacaine
- Deep soft tissue/surgical site injection (Active Comparator): A total volume of 100ml will be comprised of 60ml of 0.9% normal saline + 20ml 0.5% bupivacaine + 20ml liposomal bupivacaine will be injected into the deep soft tissue using an 18 or 20 gauge needle prior to or after prosthesis insertion
  Interventions: Drug: liposomal bupivacaine

INTERVENTIONS:
Drug: Ropivacaine — Patients will have an interscalene block under ultrasound guidance and receive .5% ropivacaine pre-operatively. Upon arrival to the Post-Operative Care Unit a continuous infusion of .5% ropivacaine will be started at 8ml/hr and increased by 2ml/hr every 15 minutes for pain score > 4 with a maximum rate of 14ml/hr. Infusion will be delivered by ON-Q Select-a-Flow pump (volume 750ml)
  Other Names: There is not another intervention involved.
  Arms: Interscalene Block
Drug: liposomal bupivacaine — A total injection volume of 100ml will be comprised of 60ml 0.9% normal saline+ 20ml .5% bupivacaine + 20ml liposomal bupivacaine will be administered into the deep tissue of the operative are with an 18 or 20 gauge needle.
  Other Names: there is not another intervention involved. Please explain to me what you are referring to.
  Arms: Deep soft tissue/surgical site injection

SUMMARY:
The purpose of the study is to determine if pain management after total shoulder arthroplasty is more efficacious with ultrasound guided, continuous Interscalene block or with local tissue infiltration with liposomal bupivacaine.

Traditionally, general anesthesia followed by narcotics has been the primary management of pain control. However, regional anesthesia in the form of an interscalene block (ISB), a perineural local anesthetic infusion, is commonly used and may more effectively control pain during and after shoulder arthroplasty, with fewer side effects than narcotics. Intraoperative benefits include better control of blood pressure and reduced need for general anesthesia and narcotics. Depending on the type of block (single shot vs. continuous) and the type of local anesthetic administered, pain relief may persist for 12-96 hours postoperatively.

However, not all patients are candidates for peripheral nerve blocks. Pre-existing pulmonary disease, previous neck surgery, cervical arthritis, neurologic disorders and obesity may preclude ISB placement. As well, interscalene blocks are not completely benign procedures. Systemic complications include clinically significant intraoperative hypotension, pneumothorax, vascular injury, cardiac arrest, respiratory failure, seizure and death. Phrenic nerve paralysis is common, although transient. Peripheral nerve injuries related to mechanical injury, medication neurotoxicity, compression or ischemia are infrequent but may be devastating. The experience and number of blocks performed by the anesthesiologist in addition to adjunctive tools, such as ultrasound and/or nerve stimulators, impacts the success of the procedure.

Continuous indwelling interscalene blocks (CISB) may provide substantial and longer pain relief, precluding the need for perioperative narcotics. Earlier discharge post procedure and better early range of motion are other purported benefits. However, premature catheter failure, catheter breakage, infection, over administration of medication and extended diaphragmatic paresis are concerns. In addition, there is a cost associated with these procedures. The anesthesiologist fee, catheter with or without elastomeric pump, local anesthetic, perioperative patient evaluation and treatment of any associated complications all must be considered.

. The development of new, long acting local anesthetics, such as liposomal bupivacaine, is potentially important in the management of perioperative pain. Liposomal bupivacaine has been approved by the US Food and Drug Administration for local infiltration for pain relief after bunionectomy and hemorrhoidectomy. This preparation increases the duration of local anesthetic action by slow release from the liposome and delays the peak plasma concentration when compared to plain bupivacaine administration. Studies have shown it to be an effective tool for postoperative pain relief with opioid sparing effects and it has also been found to have an acceptable adverse effect profile.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled study comparing post-operative pain scores, morphine sulfate equivalence consumption values, and adverse events in patients undergoing total shoulder arthroplasty with general anesthesia. Group1 will receive a pre-operative, ultrasound guided indwelling Interscalene catheter through which ropivacaine will be delivered, and Group 2 will receive intra-operative local tissue infiltration with liposomal bupivacaine. The study will enroll 80 patients, 40 in each group. Patients will be scheduled for primary conventional or reverse total shoulder arthroplasty.

Study Procedures:

Pre-Operative/ Group 1: Continuous Interscalene Block Before the patient is sedated, pre-operative pain will be assessed using the NPRS-11

* All patients to receive midazolam 0.02-0.05 mg/kg (max dose 4 mg).
* Continuous interscalene block with standardized technique:

Interscalene block under continuous ultrasound guidance with in-plane technique.

Confirmation of appropriate needle position with a bolus of D5W (3-10ml) followed by placement of interscalene catheter.

Bolus given of 30 ml 0.5% ropivacaine via the interscalene catheter with ultrasound visualization to confirm proper placement. Continuous infusion to begin immediately in PACU.

Confirmation of block by physical examination prior to proceeding to OR. If block not effective, patient to be excluded from study.

Pre-Operative/Group 2: Liposomal Bupivacaine Technique The liposomal bupivacaine will be administered by the surgeon in the OR Suite.

Pre-operative pain will be assessed using the NPRS-11 Standard shoulder arthroplasty is performed. A total injection volume of 100 cc will be comprised of 60 ml of 0.9% normal saline+ 20ml 0.5% bupivacaine + 20ml EXPAREL(liposomal bupivacaine 266mg) will be injected into the deep soft tissue using an 18 or 20 gauge needle prior to or after prosthesis insertion.

Intra Operative Management:

Once the patient is pre-medicated and the interscalene block (if appropriate) is performed, the patient is transferred to the operating room where general anesthesia (GA) is administered by standard protocol. Induction with propofol 2 to 3 mg/kg IV, 1-2 mg/kg lidocaine, and 0.5-1.0 mg/kg rocuronium. After induction and placement of the endotracheal tube, a balanced GA is maintained with Sevoflurane titrated to a minimum alveolar concentration (MAC) of 0.9 to 1.2 and muscle relaxation maintained for the needs of the procedure. If the patient's heart rate or blood pressure increases by more than 20% above pre-op value as measured in pre-op holding, an intraoperative bolus of 25 to 50 micrograms (mcg) fentanyl is administered. As per protocol, fentanyl is the only opioid used intra-operatively. At the conclusion of the surgery, muscle relaxation is reverse, the endotracheal tube is removed and the patient is transferred to PACU.

Post operative Management in PACU

Upon arrival to PACU, the patient's pain is assessed using the NPRS-11. After assessment the following medications are administered:

Continuous interscalene/Group 1:

Infusion begun immediately upon arrival at a rate of 8 ml/hr. It will be increased by 2 ml/hr every 15 minutes for a pain score >4 (≥5) with a maximum rate of 14 ml/hr. Infusion to be delivered by ON-Q Select-a-Flow pump (volume 750 ml)

* Group1 and Group 2:
* Oxycodone 5mg po every 2 hours for pain score 2-4
* Hydromorphone IV of 0.3 mg every 8 minutes PRN for pain score >4 (≥5)
* If the pain score remains >4 (≥5) after three doses, the hydromorphone dose will be increased to 0.5 mg every 8 minutes
* Patient will be switched to morphine if intolerant of hydromorphone (such as rash, pruritus, or nausea uncontrolled with ondansetron): morphine initial dose of 1.5 mg every 8 minutes and increased to 2.0 mg if needed after three doses.
* NPRS-11 pain scoring will be performed upon arrival and every 15 minutes until actual discharge from the PACU.

  5. Post-Operative Management/Patient Unit When the patient is clinically discharged from PACU by standard anesthesia protocol, they will be transferred to the post-operative patient unit. As per protocol, they will receive the following medications:
* Continuous interscalene/Group1:
* Infusion to be continued at the rate from PACU. Infusion will be increased by 2 ml/hr every 15 minutes for a pain score >4 (≥5) with a maximum rate of 14 ml/hr.
* Group 1 and Group 2:

Post-operative pain will be controlled using the following medications:

* Oxycodone 5 mg po every 2 hours for pain score 2 - 4.
* Hydromorphone IV of 0.4 mg every 30 minutes PRN for pain score >4 (≥5)
* If the pain score remains >4 (≥5) after three doses, the hydromorphone dose will be increased to 0.6-.0.8 mg every 30 minutes
* Patient will be switched to morphine if intolerant of hydromorphone (rash, pruritus, or nausea uncontrolled with ondansetron): morphine initial dose of 2 mg every 30minutes and increased to 3-4 mg if needed after three doses.
* NPRS-11 pain scoring will be performed upon arrival and at least every 4 hours.

Discharge/ Day 1-7

Patients will be discharged from the hospital when they have met the following criteria:

* Pain controlled with oral medication
* Physical Therapy (PT) will start on Post-Op Day 1. If patients are discharged the day of surgery, PT will be arranged prior to discharge.
* From a pain perspective, patients will not be discharged until pain is controlled (NPRS score of 4 or less) on oral medication. This would mean they would not be discharged home until 4 hours after their last dose of IV hydromorphone (or morphine if switched) in PACU or on the Patient Unit.
* Once discharged, patients' pain scores will be recorded twice a day. Patients will be contacted by the study nurse daily to collect the data.

Follow-Up Visits: 2Weeks, 6 Weeks, 12 Weeks

• A physical exam will be performed along with assessment of ROM and neurologic function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be between 18-75 years of age.
2. Patients must be candidates for primary total shoulder arthroplasty or reverse total shoulder arthroplasty.
3. Patients are determined by the investigator to be suitable candidates.
4. Patients must be able to understand and comply with protocol procedures.
5. Surgery must be performed at The Christ hospital Joint and Spine Center.
6. Patients must have BMI < 40 kg/m2
7. Patients must weigh a minimum of 50 kg.
8. Patients must have an American Society of Anesthesiologists(ASA) physical status I to III.

Exclusion Criteria:

1. Shoulder arthroplasty performed for an acute proximal humerus fracture.
2. Allergy or intolerance to Bupivacaine or ropivacaine.
3. Allergy to study medications: midazolam, fentanyl, hydromorphone, or oxycodone.
4. History of chronic pain, chronic narcotic use or allergy to narcotics.
5. Previous neck surgery or other anatomic abnormalities which would preclude interscalene block.
6. Failure of interscalene block placement.
7. Patients with end-stage hepatic disease.
8. Patients with end-stage renal disease requiring dialysis.
9. Patients who are pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
NPRS-11 Pain Scores | Pre-Operatively
  The Numeric Pain Rating Scale(NPRS) is an 11 point scale with 0 being no pain and 10 being extreme pain. Patients select a value that is most in line with the intensity of pain that they have experienced.
NPRS-11 Pain Scores | Upon Arrival to PACU through discharge from PACU up to 4 hours.
  The Numeric Pain Rating Scale(NPRS) is an 11 point scale with 0 being no pain and 10 being extreme pain. Patients select a value that is most in line with the intensity of pain that they have experienced. Every 15 minutes while in the Post Anesthesia Recovery Unit (PACU)
NPRS-11 Pain Scores | Upon arrival to the Patient Care Unit through Hospital Discharge up to 3 days.
  The Numeric Pain Rating Scale(NPRS) is an 11 point scale with 0 being no pain and 10 being extreme pain. Patients select a value that is most in line with the intensity of pain that they have experienced every 4 hours while in the Post-Operative patient Unit.
NPRS-11 Pain Scores | Pain scores will be recorded twice a day from hospital discharge until Post-Operative Day 7.
  The Numeric Pain Rating Scale(NPRS) is an 11 point scale with 0 being no pain and 10 being extreme pain. Patients select a value that is most in line with the intensity of pain that they have experienced.

SECONDARY OUTCOMES:
Narcotic utilization | Daily through Day 7 post-op
  Collected in morphine sulfate equivalents
Length of Stay | From Arrival to PACU through discharge form PACU up to 4 hours.
  Collected in hourly time increments
Length of Stay | From Hospital admission until hospital discharge up to 3 days.
  The amount of time the patient spent in the hospital in hourly increments.
Discharge Status | Upon patient discharge from the hospital up to 3 days.
  Will patient be discharged home or to a Skilled Nursing Facility
Procedure Cost | Through hospitalization, generally 3 days
  Record the cost of the interscalene block procedure and medication versus the cost of the liposomal bupivacaine injection.
Range of Motion | 2 weeks, 6 weeks, and 12 weeks postoperatively
  This exam will include active and passive elevation, active and passive external rotation, active and passive abduction and internal rotation.
Neurovascular Status | 2weeks, 6 weeks, and 12 weeks post-operatively
  This exam will evaluate motor function and sensation of the operative limb.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No